CLINICAL TRIAL: NCT03754907
Title: Comparing Stapled Anastomosis With Hand-sewn in Neonate With Intestinal Atresia
Brief Title: Stapled Anastomosis Versus Hand-sewn for Neonate With Intestinal Atresia
Acronym: SAVSHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, zebing Zheng, pediatric surgery, Zunyi Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zunyi Medical University
Record Dates: First submitted 2018-11-25; First posted 2018-11-27 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Intestinal Atresia; Anastomotic Complication
Keywords: stapled anastomosis; hand-sewn anastomosis; intestinal atresia; neonate
MeSH Terms: conditions — Intestinal Atresia | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stapled anastomosis group (Experimental): Following the first side-to-side anastomosis at the antimesenteric border in both intestinal limbs, the staple lines are oversewn to reinforce the crotch. Thereafter, the stapler is again fired across the joined intestinal limbs to close the enterotomies. The suture line of the side-to-side anastomosis should not overlap, and the staple lines are oversewn to reinforce the double-stapled areas.
  Interventions: Procedure: Endocutter stapler
- hand-sewn anastomosis group (Active Comparator): Patients chose HA group will performed in an end-to-end manner using absorbable suture material.
  Interventions: Procedure: suture material

INTERVENTIONS:
Procedure: Endocutter stapler — Endocutter ETS 35, ETS Flex 45 stapler, and the Echelon Flex Powered ENDOPATH Stapler with 2.5- or 3.5-mm staples (Johnson & Johnson K.K., Tokyo, Japan)
  Arms: stapled anastomosis group
Procedure: suture material — absorbable suture material is used to perform hand-sewn anastomosis in an end-to-end manner.
  Arms: hand-sewn anastomosis group

SUMMARY:
Neonatal intestinal atresia is the most difficult disease to apply stapled anastomosis. However, there are no high-quality clinical trial to verify its effectiveness. Therefore, the investigators compared the outcomes of stapled and hand-sewn anastomosis in neonate with intestinal atresia.

DETAILED DESCRIPTION:
Intestinal anastomosis in neonates with intestinal atresia has traditionally been performed using the hand-sewn end-to-end approach. After the introduction of stapled functional end-to-end anastomosis (FEEA) in neonates and infants by Powell in 1995, the procedure is gradually being accepted among pediatric surgeons. When treating intestinal atresia, great discrepancy between diameters of the proximal and distal intestine caused by disuse atrophy are often observed, which may cause difficulties and complications. To overcome size discrepancy, proficiency in performing anastomosis is required when using hand-sewn techniques. in theory, stapled functional end-to-end anastomosis does not require a special technique and does not impair the passage of intestinal contents immediately after completion because the side-to-side nature of the procedure retains the unique diameter of the target intestine and preserves patency. Stapled side-to-side functional end-to-end intestinal anastomosis is a potentially useful technique that is not affected by intestinal size discrepancy and does not require specialized surgical experience.To date, there have been a few studies about the safety and efficacy of stapled anastomosis in neonates and infants, which reported the efficacy of stapled over hand-sewn anastomosis, including shorter operative time, time to full feeding and hospitalization, and no difference in adverse outcomes between both types of anastomoses. These studies compared the clinical outcomes in neonates and infants. However,there are no high-quality clinical trials to verify its effectiveness. Therefore, the investigators compared the outcomes of stapled FEEA and hand-sewn anastomosis in neonate with intestinal atresia.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they were between 1 day and 30 days of age, and if they suffered from intestinal atresia.

Exclusion Criteria:

* These patients were complicated with intestinal perforation and peritonitis, instability of vital signs.
* Stapled anastomosis could not be performed when the intestinal lumen could not admit a 22-Fr soft catheter.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment success rate | 1 year
  Treatment success rate is defined as a patient successfully undergoing two respectively operative methods in two groups , resulting in discharge from the hospital without the need for reoperation intervention and no complication happened during a minimum follow-up of 1 year (treatment efficacy).

SECONDARY OUTCOMES:
Operative time(minute) | 1 year
  the operative time(minute) in two groups
Estimated blood loss(ml) | 1 year
  the surgeon estimated blood loss(ml) in two groups
Time to initial oral feeding | 1 year
  the time patients from operation to the first oral feeding.
Time to full oral feeding | 1 year
  the time patients from operation to the full oral feeding.
anastomotic leakage and stricture | 1year
  the incidence of complications include the anastomotic leakage and stricture between stapled anastomosis and hand-sewn anastomosis.
ileus | 1 year
  the incidence of ileus after operations 1 year in two groups
volvulus | 1 year
  the incidence of Volvulus with adhesive bands and malrotation because of anastomotic dilatation in two groups after operation 1year
reoperation | 1 year
  the incidence of complication requiring reoperation

OTHER OUTCOMES:
classification | 3 year
  counted the classification of intestinal atresia

CONTACTS AND LOCATIONS:
Overall Officials: Yuanmei Liu, Study Director — Zunyi Medical College
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

REFERENCES:
- [Background] Sato K, Uchida H, Tanaka Y, Takazawa S, Jimbo T, Deie K. Stapled intestinal anastomosis is a simple and reliable method for management of intestinal caliber discrepancy in children. Pediatr Surg Int. 2012 Sep;28(9):893-8. doi: 10.1007/s00383-012-3146-y. PMID 22864546
- [Background] Amano H, Tanaka Y, Tainaka T, Hinoki A, Kawashima H, Kakihara T, Morita K, Uchida H. The impact of body weight on stapled anastomosis in pediatric patients. J Pediatr Surg. 2018 Oct;53(10):2036-2040. doi: 10.1016/j.jpedsurg.2018.04.030. Epub 2018 Apr 26. PMID 29792281
- [Derived] Zheng Z, Jin Z, Gao M, Tang C, Gong Y, Huang L, Liu Y, Wang J. Comparison of Hand-Sewn with Stapled Anastomosis in Neonatal Intestinal Atresia Surgery: A Randomized Controlled Study. J Laparoendosc Adv Surg Tech A. 2022 Jun;32(6):696-701. doi: 10.1089/lap.2021.0714. Epub 2022 Apr 11. PMID 35404135